CLINICAL TRIAL: NCT02487446
Title: A Multi-center, Randomized, Double-blind, Double-dummy, Active Controlled, 2-period Cross-over Study to Assess the Efficacy, Safety and Tolerability of Indacaterol Maleate/Glycopyrronium Bromide Compared to Umeclidinium Bromide/Vilanterol in COPD Patients With Moderate to Severe Airflow Limitation
Brief Title: Efficacy and Safety Study of QVA149 in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2349
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Glycopyrrolate; GSK573719; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First QVA149, then Umeclidinium/vilanterol (Experimental): Participants received QVA149 27.5/12.5 ug via inhalation twice daily (b.i.d.) for 12 weeks. Then after 3 weeks washout, participants received Umeclidinium/vilanterol 62.5/25 ug via inhalation once daily for 12 weeks.
  Interventions: Drug: QVA149; Drug: Umeclidinium/vilanterol; Drug: Placebo (umeclidinium/vilanterol); Drug: Placebo (QVA149)
- First Umeclidinium/vilanterol, then QVA149 (Experimental): Participants received Umeclidinium/vilanterol 62.5/25 ug via inhalation once daily for 12 weeks. Then after 3 weeks washout, participants received QVA149 27.5/12.5 ug via inhalation twice daily (b.i.d.) for 12 weeks.
  Interventions: Drug: QVA149; Drug: Umeclidinium/vilanterol; Drug: Placebo (umeclidinium/vilanterol); Drug: Placebo (QVA149)

INTERVENTIONS:
Drug: QVA149 — QVA149 capsules for inhalation, delivered via QVA149 single dose dry powder inhaler (SDDPI)
  Other Names: Indecaterol maleate/glycopyrronium bromide
Drug: Umeclidinium/vilanterol — Umeclidinium/vilanterol for inhalation, delivered via ELLIPTA® inhaler
  Other Names: ELLIPTA®
Drug: Placebo (umeclidinium/vilanterol) — Matching Placebo to umeclidinium/vilanterol for inhalation, delivered via ELLIPTA® inhaler
Drug: Placebo (QVA149) — Matching Placebo to QVA149 capsules for inhalation, delivered via QVA149 SDDPI

SUMMARY:
The purpose of this study is to demonstrate that the efficacy of the combination product QVA149 is similar to the efficacy of the combination product umeclidinium/vilanterol on a pre-specified endpoint of FEV1 AUC0-24h while maintaining an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 yrs
* Smoking history of at least 10 pack years
* Diagnosis of stable Chronic Obstructive Pulmonary Disease (COPD) as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2015)
* Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)< 80% and ≥ 30% of the predicted normal value and post-bronchodilator FEV1/FVC (forced vital capacity) <70%
* Modified Medical Research Council questionnaire grade of 2 or higher

Exclusion Criteria:

* Patients who have had a respiratory tract infection within 4 weeks prior to Visit 1
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular co-morbid conditions
* Patients with a known history and diagnosis of alpha-1 antitrypsin deficiency
* Patients in the active phase of a supervised pulmonary rehabilitation program
* Patients contraindicated for inhaled anticholinergic agents and β2 agonists
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (55):
  - Novartis Investigative Site, Andalusia, Alabama
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Jasper, Alabama
  - Novartis Investigative Site, Multiple Locations, Alabama
  - Novartis Investigative Site, Multiple Locations, Arizona
  - Novartis Investigative Site, Tempe, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Fayetteville, Arkansas
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Rancho Mirage, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Altamonte Springs, Florida
  - Novartis Investigative Site, DeLand, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Kissimmee, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Conyers, Georgia
  - Novartis Investigative Site, Duluth, Georgia
  - Novartis Investigative Site, Meridian, Idaho
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Sunset, Louisiana
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Plymouth, Minnesota
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cornelius, North Carolina
  - Novartis Investigative Site, Gastonia, North Carolina
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Huntersville, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dublin, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Tipton, Pennsylvania
  - Novartis Investigative Site, Carrollton, Texas
  - Novartis Investigative Site, Channelview, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Lampasas, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, New Braunfels, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kerwin E, Ferguson GT, Sanjar S, Goodin T, Yadao A, Fogel R, Maitra S, Sen B, Ayers T, Banerji D. Dual Bronchodilation with Indacaterol Maleate/Glycopyrronium Bromide Compared with Umeclidinium Bromide/Vilanterol in Patients with Moderate-to-Severe COPD: Results from Two Randomized, Controlled, Cross-over Studies. Lung. 2017 Dec;195(6):739-747. doi: 10.1007/s00408-017-0055-9. Epub 2017 Oct 9. PMID 28993871

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 2 sequences in a 1:1 ratio.
Period: Period 1
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Started | 178 | 179
Completed | 165 | 171
Not Completed | 13 | 8
Not completed — Physician Decision | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol deviation | 3 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 5 | 5
Period: Washout
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Started | 165 | 171
Completed | 162 | 163
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Adverse Event | 2 | 2
Period: Period 2
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Started | 162 | 163
Completed | 154 | 158
Not Completed | 8 | 5
Not completed — Protocol deviation | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 6 | 2

BASELINE CHARACTERISTICS:
Population: Since this is a cross-over design study, all participants were randomized to receive both treatments, either in sequence QVA/UV or sequence UV/QVA. Therefore, the baseline characteristics are reported as overall participants.
Groups:
- Overall Participants: Participants received QVA149 27.5/12.5 ug via inhalation twice daily (b.i.d.) for 12 weeks and Umeclidinium/vilanterol 62.5/25 ug via inhalation once daily for 12 weeks.
Arm/Group | Overall Participants
Number analyzed (Participants) | 357
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 186

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) Area Under the Curve (AUC) 0-24h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over an entire day (AUC 0-24h). A positive change from baseline indicates improvement.
Time Frame: baseline, 0 to 24 hours post-dose at week 12
Population: The full analysis, which included all randomized patients who received at least one dose of double-blind treatment, was considered for the analysis. Only participants with a value at both baseline and the post-baseline time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- QVA149: Participants received QVA149 27.5/12.5 ug via inhalation twice daily (b.i.d.) for 12 weeks.
- Umeclidinium/Vilanterol: Participants received Umeclidinium/vilanterol 62.5/25 ug via inhalation b.i.d. for 12 weeks.
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 315 | 319
Liters | 0.2321 (0.01133) | 0.2436 (0.01130)
Statistical Analysis 1: Comparison: QVA149 vs Umeclidinium/Vilanterol; Ho: QVA149 27.5/12.5 μg b.i.d. is inferior to umeclidinium/vilanterol 62.5/25 μg q.d; Ha: QVA149 27.5/12.5 μg b.i.d. is non-inferior to umeclidinium/vilanterol 62.5/25 μg q.d; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the lower limit (LL) of the 97.5% one -sided confidence interval (CI) > -20 mL; p = 0.139, Linear Mixed Model — p-value unadjusted; Mean Difference (Net) = -0.0115, 95% CI 2-sided [-0.0269 to 0.0038], Standard Error of Mean 0.00778

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) Area Under the Curve (AUC) 0-24h
Description: as for outcome 1
Time Frame: baseline, 0 to 24 hours post-dose at week 12
Population: The full analysis, which included all randomized patients who received at least one dose of double-blind treatment, was considered for the analysis. Only participants with a value at both baseline and post-baseline time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 315 | 319
Liters | 0.2321 (0.01133) | 0.2436 (0.01130)
Statistical Analysis 1: Comparison: QVA149 vs Umeclidinium/Vilanterol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -0.0115, 95% CI 2-sided [-0.0269 to 0.0038], Standard Error of Mean 0.00778

3. Secondary Outcome: Change From Baseline in Trough FEV1 (Mean of 23h 15 Minutes and 23 h 45 Minutes Post Previous Morning Dose)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 15 minutes and 23 hours 45 minutes post-dose for each treatment
Time Frame: baseline, 23 hours 15 minutes and 23 hours 45 minutes post previous morning dose at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 309 | 310
Liters | 0.1891 (0.01070) | 0.2043 (0.01069)
Statistical Analysis 1: Comparison: QVA149 vs Umeclidinium/Vilanterol; Test type: Superiority or Other; Mean Difference (Net) = -0.0153, 95% CI 2-sided [-0.0361 to 0.0056], Standard Error of Mean 0.01062

4. Secondary Outcome: Change From Baseline in FEV1 AUC 12-24h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over 12 hours (AUC 12-24h).
Time Frame: baseline, 12 hours to 24 hours post-dose at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 312 | 316
Liters | 0.2076 (0.01159) | 0.2025 (0.01156)
Statistical Analysis 1: Comparison: QVA149 vs Umeclidinium/Vilanterol; Test type: Superiority or Other; Mean Difference (Net) = 0.0051, 95% CI 2-sided [-0.0108 to 0.0209], Standard Error of Mean 0.00806

5. Secondary Outcome: Change From Baseline in FEV1 AUC 0-12h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over 12 hours (AUC 0-12h).
Time Frame: baseline, 0 to 12 hours post-dose at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 313 | 319
Liter | 0.2543 (0.01031) | 0.2848 (0.01026)

6. Secondary Outcome: Change From Baseline in FEV1 AUC 0-4h, AUC 4-8h, AUC 8-12h, AUC 12-16h, AUC 16-20h and AUC 20-24h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over 4 hour intervals FEV1 AUC 0-4h, AUC 4-8h, AUC 8-12h, AUC 12-16h, AUC 16-20h and AUC 20-24h.
Time Frame: baseline, 12 weeks
Population: The full analysis, which included all randomized patients who received at least one dose of double-blind treatment, was considered for the analysis. Only participants with a value at both baseline and the post-baseline time points were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 341 | 340
Liter
  0-4h: number analyzed (Participants) | 312 | 319
  0-4h | 0.3223 (0.01087) | 0.3289 (0.01080)
  4-8h: number analyzed (Participants) | 311 | 317
  4-8h | 0.2399 (0.01051) | 0.2831 (0.01045)
  8-12h: number analyzed (Participants) | 308 | 315
  8-12h | 0.1911 (0.01069) | 0.2411 (0.01062)
  12-16h: number analyzed (Participants) | 309 | 315
  12-16h | 0.2594 (0.01241) | 0.2349 (0.01236)
  16-20h: number analyzed (Participants) | 308 | 312
  16-20h | 0.1914 (0.01247) | 0.1875 (0.01244)
  20-24h (n=310,314): number analyzed (Participants) | 310 | 314
  20-24h (n=310,314) | 0.1722 (0.01136) | 0.1821 (0.01133)

7. Secondary Outcome: Change From Baseline in Pre-dose Trough FEV1 (Mean of 15 Minutes and 45 Minutes Pre Morning Dose)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Pre-dose trough FEV1 was defined as the average of measurements made 15 minutes and 45 minutes pre morning dose for each treatment.
Time Frame: baseline, 15 minutes and 45 minutes pre morning dose at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 314 | 318
Liter | 0.2302 (0.01138) | 0.2450 (0.01135)

8. Secondary Outcome: QVA149 Compared to Umeclidinium/Vilanterol in Terms of Change From Baseline in FEV1 at Any Time Point
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards.
Time Frame: Day 1 (5min, 15min, 30min, hours 1, 2, 4, 8, 11h 55min, 23h 15min, 23h 45min); week 6 (-45min, -15min); week 12 (-45min, -15min, 5min, 15min, 30min, hours 1, 2, 4, 8, 11h 55min, 12h 5min, 12h 15min, 12h 30min, 13, 14, 16, 20, 23h 15min, 23h 45min)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 341 | 340
Liter
  Day 1, 5 minutes: number analyzed (Participants) | 322 | 326
  Day 1, 5 minutes | 0.1112 (0.01011) | 0.1201 (0.01007)
  Day 1, 15 minutes: number analyzed (Participants) | 320 | 319
  Day 1, 15 minutes | 0.1509 (0.01046) | 0.1682 (0.01048)
  Day 1, 30 minutes: number analyzed (Participants) | 329 | 329
  Day 1, 30 minutes | 0.1602 (0.01071) | 0.1945 (0.01073)
  Day 1, 1 hour: number analyzed (Participants) | 325 | 331
  Day 1, 1 hour | 0.1755 (0.01105) | 0.2230 (0.01100)
  Day 1, 2 hours: number analyzed (Participants) | 326 | 331
  Day 1, 2 hours | 0.1840 (0.01161) | 0.2329 (0.01157)
  Day 1, 4 hours: number analyzed (Participants) | 328 | 330
  Day 1, 4 hours | 0.1432 (0.01107) | 0.2270 (0.01105)
  Day 1, 8 hours: number analyzed (Participants) | 326 | 325
  Day 1, 8 hours | 0.0815 (0.01054) | 0.1861 (0.01056)
  Day 1, 11 hours 55 minutes: number analyzed (Participants) | 304 | 318
  Day 1, 11 hours 55 minutes | 0.0699 (0.01153) | 0.1674 (0.01138)
  Day 1, 23 hours 15 minutes: number analyzed (Participants) | 312 | 326
  Day 1, 23 hours 15 minutes | 0.1498 (0.01078) | 0.1764 (0.01063)
  Day 1, 23 hours 45 minutes: number analyzed (Participants) | 315 | 328
  Day 1, 23 hours 45 minutes | 0.1579 (0.01103) | 0.1932 (0.01090)
  Week 6, -45 minutes: number analyzed (Participants) | 317 | 319
  Week 6, -45 minutes | 0.2122 (0.01143) | 0.2469 (0.01141)
  Week 6, -15 minutes: number analyzed (Participants) | 311 | 314
  Week 6, -15 minutes | 0.2378 (0.01181) | 0.2668 (0.01179)
  Week 12, -45 minutes: number analyzed (Participants) | 311 | 314
  Week 12, -45 minutes | 0.2225 (0.01149) | 0.2378 (0.01146)
  Week 12, -15 minutes: number analyzed (Participants) | 311 | 314
  Week 12, -15 minutes | 0.2390 (0.01182) | 0.2538 (0.01179)
  Week 12, 5 minutes: number analyzed (Participants) | 308 | 310
  Week 12, 5 minutes | 0.2879 (0.01029) | 0.2831 (0.01027)
  Week 12, 15 minutes: number analyzed (Participants) | 294 | 298
  Week 12, 15 minutes | 0.3187 (0.01079) | 0.3074 (0.01074)
  Week 12, 30 minutes: number analyzed (Participants) | 301 | 312
  Week 12, 30 minutes | 0.3346 (0.01103) | 0.3258 (0.01091)
  Week 12, 1 hour: number analyzed (Participants) | 304 | 313
  Week 12, 1 hour | 0.3426 (0.01128) | 0.3334 (0.01119)
  Week 12, 2 hours: number analyzed (Participants) | 303 | 314
  Week 12, 2 hours | 0.3343 (0.01188) | 0.3445 (0.01175)
  Week 12, 4 hours: number analyzed (Participants) | 302 | 312
  Week 12, 4 hours | 0.2760 (0.01137) | 0.3137 (0.01126)
  Week 12, 8 hours: number analyzed (Participants) | 304 | 311
  Week 12, 8 hours | 0.2033 (0.01078) | 0.2545 (0.01071)
  Week 12, 11 hours 55 minutes: number analyzed (Participants) | 276 | 307
  Week 12, 11 hours 55 minutes | 0.1764 (0.01189) | 0.2311 (0.01151)
  Week 12, 12 hours 5 minutes: number analyzed (Participants) | 294 | 305
  Week 12, 12 hours 5 minutes | 0.2343 (0.01257) | 0.2218 (0.01242)
  Week 12, 12 hours 15 minutes: number analyzed (Participants) | 296 | 304
  Week 12, 12 hours 15 minutes | 0.2465 (0.01291) | 0.2324 (0.01282)
  Week 12, 12 hours 30 minutes: number analyzed (Participants) | 296 | 300
  Week 12, 12 hours 30 minutes | 0.2695 (0.01307) | 0.2350 (0.01302)
  Week 12, 13 hours: number analyzed (Participants) | 292 | 301
  Week 12, 13 hours | 0.2749 (0.01305) | 0.2448 (0.01294)
  Week 12, 14 hours: number analyzed (Participants) | 290 | 306
  Week 12, 14 hours | 0.2667 (0.01331) | 0.2355 (0.01314)
  Week 12, 16 hours: number analyzed (Participants) | 290 | 298
  Week 12, 16 hours | 0.2230 (0.01306) | 0.2197 (0.01296)
  Week 12, 20 hours: number analyzed (Participants) | 291 | 298
  Week 12, 20 hours | 0.1622 (0.01281) | 0.1629 (0.01273)
  Week 12, 23 hours 15 minutes (n=299,305): number analyzed (Participants) | 299 | 305
  Week 12, 23 hours 15 minutes (n=299,305) | 0.1791 (0.01095) | 0.1981 (0.01088)
  Week 12, 23 hours 45 minutes: number analyzed (Participants) | 300 | 303
  Week 12, 23 hours 45 minutes | 0.2048 (0.01122) | 0.2117 (0.01118)

9. Secondary Outcome: QVA149 Compared to Umeclidinium/Vilanterol in Terms of Change From Baseline in Forced Vital Capacity (FVC) at Any Time Point
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards.
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QVA149 | Umeclidinium/Vilanterol
Number analyzed (Participants) | 341 | 340
Liter
  Day 1, 5 minutes: number analyzed (Participants) | 322 | 326
  Day 1, 5 minutes | 0.2177 (0.01732) | 0.2218 (0.01726)
  Day 1, 15 minutes: number analyzed (Participants) | 320 | 319
  Day 1, 15 minutes | 0.2566 (0.01818) | 0.2927 (0.01821)
  Day 1, 30 minutes: number analyzed (Participants) | 329 | 329
  Day 1, 30 minutes | 0.2811 (0.01846) | 0.3325 (0.01849)
  Day 1, 1 hour: number analyzed (Participants) | 325 | 331
  Day 1, 1 hour | 0.2944 (0.01912) | 0.3534 (0.01904)
  Day 1, 2 hours: number analyzed (Participants) | 326 | 331
  Day 1, 2 hours | 0.3109 (0.01966) | 0.3687 (0.01960)
  Day 1, 4 hours: number analyzed (Participants) | 328 | 330
  Day 1, 4 hours | 0.2788 (0.04347) | 0.4237 (0.04339)
  Day 1, 8 hours: number analyzed (Participants) | 326 | 325
  Day 1, 8 hours | 0.1681 (0.01816) | 0.3237 (0.01818)
  Day 1, 11 hours 55 minutes: number analyzed (Participants) | 304 | 318
  Day 1, 11 hours 55 minutes | 0.1406 (0.01915) | 0.2910 (0.01889)
  Day 1, 23 hours 15 minutes: number analyzed (Participants) | 312 | 326
  Day 1, 23 hours 15 minutes | 0.2565 (0.01777) | 0.2747 (0.01753)
  Day 1, 23 hours 45 minutes: number analyzed (Participants) | 315 | 328
  Day 1, 23 hours 45 minutes | 0.2737 (0.01903) | 0.3001 (0.01883)
  Week 6, -45 minutes: number analyzed (Participants) | 317 | 319
  Week 6, -45 minutes | 0.2914 (0.01853) | 0.3513 (0.01851)
  Week 6, -15 minutes: number analyzed (Participants) | 311 | 314
  Week 6, -15 minutes | 0.3390 (0.01922) | 0.3732 (0.01919)
  Week 12, -45 minutes: number analyzed (Participants) | 311 | 314
  Week 12, -45 minutes | 0.3044 (0.01864) | 0.3442 (0.01859)
  Week 12, -15 minutes: number analyzed (Participants) | 311 | 314
  Week 12, -15 minutes | 0.3344 (0.01923) | 0.3566 (0.01919)
  Week 12, 5 minutes: number analyzed (Participants) | 308 | 310
  Week 12, 5 minutes | 0.3960 (0.01760) | 0.3861 (0.01756)
  Week 12, 15 minutes: number analyzed (Participants) | 294 | 298
  Week 12, 15 minutes | 0.4378 (0.01865) | 0.4169 (0.01857)
  Week 12, 30 minutes: number analyzed (Participants) | 301 | 312
  Week 12, 30 minutes | 0.4602 (0.01892) | 0.4480 (0.01875)
  Week 12, 1 hour: number analyzed (Participants) | 304 | 313
  Week 12, 1 hour | 0.4649 (0.01948) | 0.4647 (0.01934)
  Week 12, 2 hours: number analyzed (Participants) | 303 | 314
  Week 12, 2 hours | 0.4405 (0.02006) | 0.4853 (0.01987)
  Week 12, 4 hours: number analyzed (Participants) | 302 | 312
  Week 12, 4 hours | 0.3872 (0.04490) | 0.4343 (0.04435)
  Week 12, 8 hours: number analyzed (Participants) | 304 | 311
  Week 12, 8 hours | 0.2714 (0.01856) | 0.3555 (0.01844)
  Week 12, 11 hours 55 minutes: number analyzed (Participants) | 276 | 307
  Week 12, 11 hours 55 minutes | 0.2306 (0.01977) | 0.3231 (0.01911)
  Week 12, 12 hours 5 minutes (n=294,305): number analyzed (Participants) | 294 | 305
  Week 12, 12 hours 5 minutes (n=294,305) | 0.3455 (0.02063) | 0.3112 (0.02038)
  Week 12, 12 hours 15 minutes: number analyzed (Participants) | 296 | 304
  Week 12, 12 hours 15 minutes | 0.3409 (0.02086) | 0.3235 (0.02070)
  Week 12, 12 hours 30 minutes: number analyzed (Participants) | 296 | 300
  Week 12, 12 hours 30 minutes | 0.3688 (0.02196) | 0.3326 (0.02187)
  Week 12, 13 hours: number analyzed (Participants) | 292 | 301
  Week 12, 13 hours | 0.3760 (0.02123) | 0.3361 (0.02104)
  Week 12, 14 hours: number analyzed (Participants) | 290 | 306
  Week 12, 14 hours | 0.3681 (0.02192) | 0.3371 (0.02162)
  Week 12, 16 hours: number analyzed (Participants) | 290 | 298
  Week 12, 16 hours | 0.3129 (0.02205) | 0.3279 (0.02189)
  Week 12, 20 hours: number analyzed (Participants) | 291 | 298
  Week 12, 20 hours | 0.2175 (0.02180) | 0.2353 (0.02167)
  Week 12, 23 hours 15 minutes: number analyzed (Participants) | 299 | 305
  Week 12, 23 hours 15 minutes | 0.2237 (0.01804) | 0.2750 (0.01792)
  Week 12, 23 hours 45 minutes (n=300,303): number analyzed (Participants) | 300 | 303
  Week 12, 23 hours 45 minutes (n=300,303) | 0.2607 (0.01935) | 0.2728 (0.01928)

ADVERSE EVENTS:
Description: Since this is a cross-over design study, all patients were randomized to receive both treatments, either in sequence QVA/UV or sequence UV/QVA. The number of patients on each treatment does not add up to the total number of patients.
Groups:
- All Patients: All Patients
Arm/Group | QVA149 | Umeclidinium/Vilanterol | All Patients
Serious Adverse Events (participants affected / at risk) | 13/341 | 21/340 | 33/356
Other Adverse Events (participants affected / at risk) | 85/341 | 104/340 | 161/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=341) | Umeclidinium/Vilanterol (N=340) | All Patients (N=356)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 5 | 6
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=341) | Umeclidinium/Vilanterol (N=340) | All Patients (N=356)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 4
Nausea (Gastrointestinal disorders) | 3 | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4
Fatigue (General disorders) | 2 | 2 | 4
Bronchitis (Infections and infestations) | 5 | 11 | 15
Lower respiratory tract infection (Infections and infestations) | 3 | 3 | 6
Nasopharyngitis (Infections and infestations) | 19 | 12 | 28
Sinusitis (Infections and infestations) | 4 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 11 | 16
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 4 | 5
Viral upper respiratory tract infection (Infections and infestations) | 4 | 6 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Headache (Nervous system disorders) | 3 | 5 | 8
Anxiety (Psychiatric disorders) | 2 | 3 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 36 | 50 | 76
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 14
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Hypertension (Vascular disorders) | 3 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.